CLINICAL TRIAL: NCT00813449
Title: Multicenter, Double-blinding, Randomized Controlled, Phase II Clinical Trial on Combined Chemotherapy of Endostar (Recombinant Human Endostatin) for Untreated Patients With Advanced Melanoma
Brief Title: Safety Study of Combined Chemotherapy and Endostar to Untreated Patients With Advanced Melanoma
Acronym: melanoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Simcere Pharmaceutical Co., Ltd (Other)
Responsible Party: Guo Jun, Expert Committee for Melanoma of CSCO
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: simcere001; simcere0801
Record Dates: First submitted 2008-12-19; First posted 2008-12-23 (Estimated); Last update posted 2009-12-08 (Estimated); Status verified 2009-11

CONDITIONS: Advanced Melanoma; Untreated Patients
Keywords: Endostar; advanced melanoma; combined chemotherapy
MeSH Terms: interventions — Dacarbazine; endostar protein; Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Experimental group : Endostar combined with dacarbazine
  Interventions: Drug: dacarbazine plus Endostar (Experimental group)
- 2 (Placebo Comparator): Control group : Dacarbazine combined with placebo
  Interventions: Drug: dacarbazine plus placebo (control group)

INTERVENTIONS:
Drug: dacarbazine plus Endostar (Experimental group) — dacarbazine plus Endostar
  Other Names: dacarbazine plus Endostar
  Arms: A
Drug: dacarbazine plus placebo (control group) — dacarbazine plus placebo
  Other Names: dacarbazine plus placebo
  Arms: 2

SUMMARY:
Multicenter, double-blinding, randomized controlled, phase II clinical trial on combined chemotherapy of Endostar (Recombinant Human Endostatin) for untreated patients with advanced melanoma, To compare the efficacy and safety of Endostar combined with Dacarbazine and monotherapy of Dacarbazine for advanced melanoma

DETAILED DESCRIPTION:
Dacarbazine (DTIC) has been approved for treating metastatic melanoma in the 1970s, and as a single agent gives a response rate of about 20%. There have been efforts to ameliorate this poor result by using DTIC in different combinations without a significant improvement. In addition, new studies with melanoma cells in vitro show that DTIC combination with Endostar, suggesting a potential clinical benefit from the concomitant treatment of DTIC and antiangiogenesis therapy. Endostar is a wild spectrum and safe antiangiogenesis factor which could suppress almost 65 kinds of tumor mass in animal models and affect about 12 percent human genome. The purpose of this study is to determine whether a combination therapy of endostar and DTIC is safe and can increase response rate and progression-free survival in patients (pts) with metastatic melanoma. We will evaluate the efficacy and safety of the Endostar plus DTIC and hope provide a new hope for the advanced melanoma patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old, males or females;
2. Untreated patients with advanced melanoma confirmed by histopathology or cytology;
3. With tumor foci that can be evaluated by CT or MRI; at least one diameter ≥ 1 cm (including metastatic lymph nodes, diameter ≥ 1 cm confirmed by CT scan); or superficial focus ≥ 2 cm (confirmed by photos with calibration);
4. No contraindication for chemotherapy, with normal peripheral hemogram, renal and hepatic function: Peripheral hemogram: WBC≥4.0×109/L，PLT≥80×109/L，Hgb≥90g/L； Renal function: serum BUN and creatinine ≤2.5×UNL; Hepatic function: transaminase≤2.5×UNL, or ≤5×UNL in patients with liver metastasis;
5. Karnofsky performance scale≥70 (appendix 1); expected survival time≥3 months;
6. Patients are voluntary to participate and sign the informed contents.

Exclusion Criteria:

1. Pregnant or breast-feeding females; or females who have reproductive ability but do not take contraception method;
2. With severe acute infection uncontrolled; purulent or chronic infection with wounds difficult to recover;
3. With history of severe heart diseases, including congestive heart failure, uncontrolled arrhythmia with high risk, unstable angina pectoris, myocardial infarction, severe cardiac valvular diseases and refractory hypertension;
4. Have been treated by dacarbazine or dacarbazine included combination chemotherapy;
5. Patients with uncontrolled neurological, mental disease or psychosis, patients with poor compliance that cannot coordinate the therapy or describe the treatment response;
6. Uncontrolled brain metastasis patients with obvious manifestations of intracranial hypertension or neurological and mental disorders;
7. Allergic to any drug in the trial;
8. Patients with a second tumor;
9. Patients participating in other clinical trials;
10. Other conditions that are regarded for exclusion by the trialists

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2008-08; Primary Completion 2010-08 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival time , Total survival time | 2010.8

SECONDARY OUTCOMES:
Tumor response rate , Disease controlled rate and adverse effects | 2009.8

CONTACTS AND LOCATIONS:
Overall Officials: Guo Jun, PI, Principal Investigator — Expert Committee for Melanoma of CSCO
Locations (1):
- Beijing tumor hospital, Beijing, Beijing Municipality, China

REFERENCES:
- See also: Related Info — http://www.bjcancer.org/